CLINICAL TRIAL: NCT04935411
Title: Russian Registry of Patients With Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: Russian Registry of Patients With nAMD
Status: Terminated | Type: Observational
Why Stopped: Enough participants were included, which made it possible to answer the objectives of the study.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258ARU01
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration; nAMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- nAMD patients: patients diagnosed with Neovascular Age-Related Macular Degeneration
  Interventions: Other: nAMD

INTERVENTIONS:
Other: nAMD — patients diagnosed with Neovascular Age-Related Macular Degeneration

SUMMARY:
A three-year, non-randomized, observational, multicenter prospective nAMD study - patient registry.

DETAILED DESCRIPTION:
The registry is a structured system which uses observational study methods for systematic collection of data on health condition in the specific patient population.

Real world clinical practice data will be collected. Patients will not undergo any additional examinations or procedures that are outside of the standard clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Age > to 18 years
* Male or female patients diagnosed with nAMD (with or without previous treatment for nAMD including but not limited to PDT, laser coagulation, vitamins, retinolamine, emoxipine, anti-VEGF therapy or any surgery for nAMD).
* Willing and able to provide informed written consent personally or by legal proxy

Exclusion Criteria:

* The patient does not meet the inclusion criteria;
* The patient is simultaneously participating in a different nAMD therapy study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Neovascular Age-Related Macular Degeneration in Russia
Sampling Method: Non-Probability Sample
Enrollment: 2665 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Number of patients by gender | Baseline
  Number of patients by gender to be provided
Age at the diagnosis | Baseline
  Age at the diagnosis to be provided
Percentage of patients with comorbidities and concomitant procedures and medications | Baseline
  Percentage of patients with systemic and ophthalmic comorbidities and percentage of patients with concomitant procedures and medications to be provided
Patients with unilateral or bilateral disease | Baseline
  Percentage of patients with unilateral or bilateral disease
Time from diagnosis to entry to the registry | Baseline
  Mean time from diagnosis to entry to the registry to be presented
Social Characteristics (Working and Disability status) | Baseline
  Working status (number of patients that work/does not work, with age-related pension, disability pension).
  Disability status (number of patients established/not established, removed, disability group, whether AMD is the main reason for disability)
Visual acuity | Baseline, up to 2 years
  Changes in visual acuity assessed by Sivcev-Golovin's table (The table consists of two parts with 12 rows each, representing visual acuity values between 0.1 and 2.0.) or Snellen equivalent
Presence of edema and/or neuroepithelium detachment and/or pigment epithelium detachment | Baseline, Up to 2 years
  Presence of edema and/or neuroepithelium detachment and/or pigment epithelium detachment. (yes/no)
Presence of macular atrophy | Baseline, Up to 2 years
  Presence of macular atrophy (with or without foveal involvement) (yes/no)
Central retinal thickness | Baseline, Up to 2 years
  Central retinal thickness to be measured with OCT (optical coherent tomography)
Fluid type | Baseline, Up to 2 years
  Type of the fluid assessed by optical coherence tomography and defined as follows: intraretinal fluid (IRF), subretinal fluid (SRF), fluid under repinal pigment epithelium (sub-RPE)
Indication for intravitreal anti-VEGF therapy | Baseline, Up to 2 years
  Indication for intravitreal anti-VEGF therapy to be collected

SECONDARY OUTCOMES:
Type of prescribed therapy | Up to 2 years
  Type of prescribed therapy (anti-VEGF, PDT, laser coagulation, retinolamine, emoxipine, etc.)
Percentage of patients with prescription of anti-VEGF drugs | Up to 2 years
  Percentage of patients with prescription of anti-VEGF drugs to be collected
Time from diagnosis to the therapy initiation | Up to 2 years
  Mean time from the diagnosis to the initiation of any therapy for nAMD
Time from diagnosis to anti-VEGF injection | Up to 2 years
  Mean time from the diagnosis to the first anti-VEGF injection
Number of visits per year | Up to 2 years
  Number of visits per year to be collected
Number of anti-VEGF injections per year | Up to 2 years
  Number of anti-VEGF injections to be collected
Number of Optical coherence tomography (OCTs) done per year | Up to 2 years
  Number of OCTs done per year to be collected
Rate of treatment discontinuation | Up to 2 years
  Rate of treatment discontinuation
Reasons for treatment discontinuation | Up to 2 years
  Reasons for treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No